CLINICAL TRIAL: NCT02552992
Title: Yoga for Chronic Low Back Pain and Its Mechanism of Action: Impact of Strength and Stretch (YoMA II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSFCHR14-14148
Record Dates: First submitted 2015-08-18; First posted 2015-09-17 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Classes (Experimental): Study Participants will receive: 12 weekly yoga classes, a book and a home practice audio recording.
  Interventions: Behavioral: Yoga
- Self-Directed Mind-Body Program (Active Comparator): Study Participants will receive: The Back Pain Helpbook, a mind-body self-care program for better living.
  Interventions: Behavioral: Self-Directed Mind-Body Program

INTERVENTIONS:
Behavioral: Yoga
  Arms: Yoga Classes
Behavioral: Self-Directed Mind-Body Program
  Arms: Self-Directed Mind-Body Program

SUMMARY:
This study is a pilot, randomized controlled trial to provide feasibility and conduct preliminary analyses on physical (strength and stretch) mechanisms associated with a yoga intervention for non-specific chronic low back pain (cLBP). Recent large-scale trials have demonstrated the efficacy of a yoga intervention for cLBP however, many types of yoga classes are available to the public and a specialized yoga protocol for individuals with cLBP is needed. This study's goal is to quantify trunk strength and flexibility to better understand how these potential physical mechanisms specifically lead to improvement in pain-related outcomes including pain and disability. This knowledge will be used to design a large scale trial of mechanisms of yoga for cLBP. For this pilot study, 40 participants will be randomized to either a yoga intervention (N=20) or to a usual care group (N=20) that will receive The Back Pain Helpbook, a mind-body self-care program for better living. The yoga intervention will be offered weekly yoga classes and instructional materials will be provided for home practice.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain lasting > 6 months
* Back pain that is rated at least 3 on a numeric pain rating scale that ranges from 0 to 10 (0-no pain, 10 worst pain imaginable).
* English language fluency

Exclusion Criteria:

* BMI > 40
* Inability to provide informed consent
* Recent diagnosis of abdominal aneurism
* Recent diagnosis of metastatic cancer
* Recent diagnosis of discitis
* Recent diagnosis of disk disease
* Recent diagnosis of spinal stenosis
* Recent diagnosis of spondylolisthesis
* Recent diagnosis of infectious cause of back pain
* Recent diagnosis of fracture of vertebra
* Recent diagnosis of Fibromyalgia
* Recent diagnosis of rheumatoid arthritis
* Recent diagnosis of ankylosing spondylitis
* Recent diagnosis of paralysis
* Pregnancy
* Prior or planned back surgery
* Blindness or severe vision problems
* Deafness or severe hearing problems
* Bipolar or manic depression and not taking medication
* Major depression
* Psychoses (major)
* a substance abuse condition
* Dementia
* Unable to get up and down from the floor
* Involvement in a lawsuit related to back pain
* Lack of transportation
* Other disabling chronic conditions (e.g., disabling heart or lung disease, diabetic neuropathy, receiving treatment for hepatitis)
* Currently (within the past 3 months) using yoga classes for more than 15 minutes per week
* Inability to be contacted by phone or email
* no computer access
* schedule does not allow for participation in classes/home practice
* planning to move out of town or take a long vacation during the period of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Roland Morris Disability Questionnaire | 6 months

SECONDARY OUTCOMES:
Change in Numeric Rating Scale for Pain | 6 months
Change in Pain Medication Usage Survey | 6 months

OTHER OUTCOMES:
Change in Strength testing (Biodex Dynamometer) | 6 months
Change in Trunk flexibility (sit-and-reach) testing | 6 months
Change in Lateral flexion (goniometer) testing | 6 months
Change in Pain Catastrophizing Scale | 6 months
Change in Multidimensional Assessment of Interoceptive Awareness | 6 months